CLINICAL TRIAL: NCT01360333
Title: Oral Fluid: Absorption and Expansion of the Blood Volume
Brief Title: Oral Fluid Volume Expansion
Acronym: OFVEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Joachim Zdolsek, MD, PhD, University Hospital, Linkoeping
Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: OFVEX
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Dehydration; Hydration
Keywords: Dehydration; Hydration
MeSH Terms: conditions — Dehydration | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tap water, sodium chloride, carbohydrate rich fluid (Other)
  Interventions: Other: tap water, sodium chloride, carbohydrate rich fluid

INTERVENTIONS:
Other: tap water, sodium chloride, carbohydrate rich fluid — Ingestion of three different fluids at three different occasions separated by at least one week, A, Tap water. B. Sodium Chloride. C. Carbohydrate rich fluid.

SUMMARY:
When subjected to fluid loss or fluid deficiency irrespective of disease or environmental factors it is discussed how to rehydrate or how to hydrate prophylactic.

In medical care it is common to give infusions. However it has increasingly become common to hydrate the patient through the mouth even early after bowel surgery. Moreover it is more simple to provide energy the natural way.

Which fluid to give, depends on several factors such as possibility to drink, the volume and emptying of the stomach as well as the fluid absorption in the bowel.

The provided fluid can also influence this process depending on temperature, osmolality/tonicity and composition (carbohydrates or salts).

In this study we wish to study the speed with which the provided fluid is absorbed by the bowels and how fast the fluid is distributed to the different body compartments depending on it's composition.

The three fluids will be either tap water, high sodium chloride and a carbohydrate rich fluid.

DETAILED DESCRIPTION:
The healthy volunteer starts the study by voiding. Then he/she lies down for 30 minutes. A blood sample is drawn and thereafter the healthy volunteer ingests one of the three fluids. Blood samples are drawn 10 times during the following two hours. Finally the healthy volunteer is asked to void and the voided urine is measured. The hemoglobin concentrations are used to calculate the blood volume expansion with volume kinetic methods.

The process is repeated another two times with the two remaining fluids.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer
* 18 to 50 years old

Exclusion Criteria:

* medication
* any chronical disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
change in hydration | 2.5 hours
  volume kinetics: calculation from hemoglobin variations

SECONDARY OUTCOMES:
fluid kinetic effects of oral carbohydrates | 2.5 hours
  Electrolytes and blod glucose will be measured to se how much these are affected by the glucose upptake.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Zdolsek, MD, PhD, Principal Investigator — University Hospital, Linköping, Sweden
Locations (1):
- Intensive Care Unit, University Hospital, Linköping, Sweden

REFERENCES:
- [Derived] Hahn RG, Wuethrich PY, Zdolsek JH. Can perioperative hemodilution be monitored with non-invasive measurement of blood hemoglobin? BMC Anesthesiol. 2021 May 6;21(1):138. doi: 10.1186/s12871-021-01351-4. PMID 33957864
- [Derived] Zdolsek J, Metander A, Hahn R. Volume kinetic evaluation of fluid turnover after oral intake of tap water, lemonade and saline in volunteers. BMC Sports Sci Med Rehabil. 2016 Jul 28;8:22. doi: 10.1186/s13102-016-0045-x. eCollection 2016. PMID 27471593